CLINICAL TRIAL: NCT04977206
Title: Engaging Patients in Mutual Goal-Setting in Hospitalized Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marquette University (Other)
Collaborators: Froedtert Hospital (Other)
Responsible Party: Principal Investigator, Teresa Jerofke-Owen, Assistant Nursing Professor, Marquette University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HR-3725
Record Dates: First submitted 2021-06-22; First posted 2021-07-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Goals

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention (No Intervention): Patients receiving usual care
- Intervention (Experimental): Patient's receiving care following nurse education on mutual goal-setting
  Interventions: Other: Mutual Goal-Setting Education

INTERVENTIONS:
Other: Mutual Goal-Setting Education — Nurses will receive both written and verbal instruction on mutual goal-setting with patients using SMART methodology
  Arms: Intervention

SUMMARY:
Mutual goal setting and action planning in patients with long-term conditions in outpatient settings is associated with favorable effects on measures of physical health, psychological health, subjective health status, self-management self-efficacy levels, activation levels, and perceived empowerment. The purpose of this study is to examine the impact of an educational intervention delivered to the staff nurses of two surgical units on how to engage patients in mutual goal-setting in the acute care setting. Staff nurses from two 32-bed surgical units will be scheduled to attend an hour-long educational intervention. A total of 630 chart audits will be conducted one month prior and one and three months following the intervention per unit, to examine the number of patients with a daily goal recorded in the prior 24 hours and the quality of the recorded goal using the SMART-GEM. The self-efficacy of engaging in mutual goal-setting with patients will be examined by asking nurses to complete the Appraisal Inventory Tool (AIT) prior to and immediately following the intervention. The patient experience of engaging in mutual goal-setting will be examined by having a total of 165 patients complete the Patient Experience of Mutual Goal-Setting Tool (PEMGST) one month prior to the intervention and one and three months following the intervention on each of the two units.

ELIGIBILITY:
Inclusion Criteria

* At least 18 years of age or older
* Must be alert and oriented to person, place, and time
* Inpatient on one of two included units

Exclusion Criteria

* Less than 24 hour length of stay
* Non English-speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of charts reviewed with an individualized goal recorded in the electronic health record | Over the course of one month before delivery of education intervention and one and three months post delivery of intervention
  percentage of charts reviewed with individualized goals recorded in their electronic health record

SECONDARY OUTCOMES:
Change in quality of goals as measured by the SMART-GEM. | Over the course of one month before delivery of education intervention and one and three months post delivery of intervention
  Quality of charted individualized goals using talhe SMART-GEM tool. The SMART-GEM (Bowman, Mogensen, Marsland, & Lannin, 2015) is an objective tool that can be used to score the quality of a SMART goal. The interrater agreement on total scores was very good (ICC=.0895, 95% CI = .743 to .986, p=.001) with excellent internal consistency (alpha = .995).
Change in patient experience with mutual goal-setting using the Patient Experience of Mutual Goal-Setting Tool. | Over the course of one month before delivery of educational intervention and one and three months post delivery of intervention
  Patient experience with mutual goal setting using the Patient Experience of Mutual Goal-Setting Tool, a 5-item survey created by PI to measure the patient experience of mutual goal-setting (involvement, satisfaction, knowledge, feeling heard, achievement of goals). Questions are on a 6-point Likert scale, with higher scores indicating a more favorable experience.
Change in nurse self-efficacy participating in mutual goal-setting with patients pre and post-intervention using the Appraisal Inventory Tool. | Immediately before starting the educational intervention and immediately following the conclusion of the educational intervention
  Nurse self-efficacy participating in mutual goal-setting with patients. The Appraisal Inventory Tool is a 5-item survey created by PI to measure nurse self-efficacy for mutual goal-setting using Bandura's (2006) guidelines. The items use an 11-point Likert scale, and higher scores indicate a higher self-efficacy score

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Memorial Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jerofke-Owen TA, Opper K, Beiler J, Singh M. An Educational Intervention on Mutual Goal Setting for Hospital Nurses: A Mixed-Methods Study. West J Nurs Res. 2026 Jan;48(1):4-14. doi: 10.1177/01939459251384711. Epub 2025 Nov 5. PMID 41190497